CLINICAL TRIAL: NCT02365077
Title: Genome-wide Association Study Identified Susceptibility Loci for Glucocorticoid-induced Femur Head Necrosis in the Chinese Population
Brief Title: GWAS Identified Susceptibility Loci for Glucocorticoid-induced FHN in the Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, xjpfW, Chief in Department of Dermatology, Xijing Hospital
Other Study IDs: CUP2015D001
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Femur Head Necrosis; Adverse Effect of Glucocorticoids and Synthetic Analogues
Keywords: Adverse Effect of Glucocorticoids; Femur Head Necrosis; Susceptibility; GWAS
MeSH Terms: conditions — Femur Head Necrosis; Disease Susceptibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — We will collect 4ml whole blood samples under the consent of patient and extract the genome from the samples. During the process the blood samples will be collected strickly according the international guide clinical blood specimen collection.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: The patients of necrosis group was defined by a history of taking 1800 mg prednisolone or an equivalent over 4 week without the symptom of femur head necrosis after 1 year.
- Necrosis: The patients of necrosis group was defined by a history of taking 1800 mg prednisolone or an equivalent over 4 week with the diagnosis of femur head necrosis.

SUMMARY:
This is a observation clinical trial. We are collecting the patients with glucocorticoid. They were divided into the experiment group (with femur head necrosis) and control group (without femur head necrosis).Then, we will analyse the patients' genome with genome-wide association study (GWAS). Our purpose is to find susceptibility loci for glucocorticoid-induced femur head necrosis in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given the written informed consent voluntarily;
2. Male or female between 18~60 years;
3. Candidate is clinically diagnosed as avascular osteonecrosis of the femoral head (ONFH), in reference to the diagnostic criteria set forth by Experts' Consensus on the Diagnosis and Treatment of Osteonecrosis of the Femoral Head in Adults (edition 2012);
4. Patient with history of glucocorticoid therapy, in form of oral, muscular or vascular administration, should have total dose equivalent to ≧2000 mg of Prednisone, and maintain on that dose for ≦3 months.

Exclusion Criteria:

1. Subject is not in conformity with diagnostic criteria for ONFH;
2. Patient has a history of trauma in the lower limbs or pelvis;
3. Prolonged addiction to alcohol;
4. Concurrent with renal failure, organ transplant, graft versus host disease, inflammatory bowel disease, HIV infection or leukemia;
5. Patient with familial idiopathic ONFH;
6. Subject suffers from a fatal disease, with life expectancy < 2 months;
7. Woman of child-bearing potential, who is pregnant, in preparation of pregnancy or breast-feeding during the study period;
8. Other patients deemed ineligible at the discretion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients coming from the Department of Dermatology Xijing Hospital, Fourth Military Medical University Xi'an, China
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucocorticoid-induced femur head necrosis | 1 year
  Hip joint MRI for the patients with a history of taking 1800 mg prednisolone or an equivalent over 4 week.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospitial, Xi'an, Shaanxi, China